CLINICAL TRIAL: NCT06710522
Title: COMPARISON OF OXIDANT-ANTIOXIDANT LEVELS WITH STRESS HORMONES IN SPINAL ANESTHESIA AND GENERAL ANESTHESIA IN LAPAROSCOPIC TUBE LIGATION
Acronym: LAP TUBE LİG
Status: Enrolling by invitation | Type: Observational
Sponsor: KADİR TEOMAN (Other Government)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor-Investigator, KADİR TEOMAN, Specialist, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Other Study IDs: AEŞH-EK1-2023-478
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Laparoscopic Surgery
Keywords: spinal anesthesia; general anesthesia; cortisol; acth; native thiol; total thiol; disulfide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS UNDERGOING LAPAROSCOPIC TUBA LIGATION SURGERY: COMPARISON OF PATIENTS UNDERGOING GENERAL AND SPINAL ANESTHESIA AS ANESTHESIA METHODS IN LAPAROSCOPIC TUBE LIGATION SURGERY

SUMMARY:
The aim of this observational study is to investigate the effect of anesthesia method applied in laparoscopic tubal ligation on stress factors in women aged 15-45. The main question it aims to answer is:

Do spinal anesthesia and general anesthesia applied during laparoscopic tubal ligation surgery cause a change in the body's stress hormones? Do patients who undergo spinal anesthesia produce less oxidant-antioxidant than patients who undergo general anesthesia? Patients will answer the State and Trait Anxiety Scale questions before the operation

DETAILED DESCRIPTION:
Laparoscopic procedures are usually performed as day surgery. General and regional anesthesia; It is used successfully and safely when care is taken in the use of short-acting drugs, ensuring cardiovascular stability, rapid recovery and mobilization, postoperative nausea, vomiting and pain treatment.

Although the common procedure in laparoscopic surgeries is surgery under general anesthesia, it has been reported that regional anesthesia methods can be used safely within certain limits.

Regional anesthesia; It is advantageous due to rapid recovery, less nausea and vomiting and postoperative pain, short hospitalization, reduced cost, increased patient satisfaction, early diagnosis of complications and less hemodynamic changes. General anesthesia complications such as sore throat, muscle pain and airway trauma are not observed.

There are some limitations when regional anesthesia methods are applied in laparoscopic surgeries. Problems in the operating room cause the patient's anxiety, pain and discomfort to increase, causing the need for intravenous sedation support. Pneumoperitoneum effect may cause sedation, hypoventilation and decrease in arterial oxygen saturation.

One of the indications for regional anesthesia is laparoscopic tubal ligation. Procedures requiring many puncture points, important organ manipulations, steep inclination of the operating table, development of pneumoperitoneum make it difficult for the patient to breathe spontaneously and regional anesthesia should not be applied in these cases.

Spinal anesthesia is the simplest and most reliable regional anesthesia technique. Spinal anesthesia, which is a primary technique for laparoscopic gynecology, has many advantages over general anesthesia.

The patient position depends on the area to be operated on. In gynecological procedures, the Trendelenburg position is applied for the pelvic organs. In laparoscopic surgeries, the operator must be experienced in order to apply spinal anesthesia. Trendelenburg position may cause spinal block to spread to the head, increase sympathetic block, bradycardia and hypotension. In rare cases, intubation material and general anesthesia devices should be immediately available to ensure deep hypotension and respiratory continuity.

Regional anesthesia has advantages such as minimal effect on the respiratory system and prevention of the spread of pathogens related to intubation to the lower respiratory system.

Reduced thromboembolic complications and reduced surgical stress response. By using regional anesthesia techniques, aerosol-generating procedures can be avoided with less risk for healthcare personnel.

Low-dose spinal anesthesia is a good alternative to general anesthesia with desflurane in outpatient gynecological surgeries. Postoperative pain and cost are less in spinal anesthesia, while recovery is faster. When compared to general anesthesia with propofol total intravenous infusion, recovery time was found to be shorter in low-dose spinal anesthesia. With the development of gasless laparoscopy and microlaparoscopy techniques, the place of spinal anesthesia in laparoscopies will increase over time.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II Women aged 18-45 Patients undergoing laparoscopic tubal ligation

Exclusion Criteria:

* Patients with psychiatric illness, Patients who developed complications during laparoscopy, Patients who converted from spinal anesthesia to general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female Adults Patients
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
kortizol-acth levels | from december 2024 to january 2025
  Determination of differences in cortisol and ACTH hormones in patients who underwent bilateral tubal ligation with spinal anesthesia compared to patients who underwent bilateral tubal ligation with general anesthesia.
oxidant-antioxidan levels | from december 2024 to january 2025
  Determination of differences in oxidant-antioxidant values in patients who underwent bilateral tubal ligation with spinal anesthesia compared to patients who underwent bilateral tubal ligation with general anesthesia.

SECONDARY OUTCOMES:
Evaluation of patient and surgical satisfaction | from january 2025 to february 2025
  Evaluation of patient and surgical satisfaction in patients undergoing bilateral tubal ligation with spinal anesthesia and in patients undergoing bilateral tubal ligation with general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: KADİR TEOMAN ETİKCAN, MEDİCAL DOCTOR, Principal Investigator — ANKARA ETLİK CİTY HOSPİTAL
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Major AL, Jumaniyazov K, Yusupova S, Jabbarov R, Saidmamatov O, Mayboroda-Major I. Laparoscopy in Gynecologic and Abdominal Surgery in Regional (Spinal, Peridural) Anesthesia, the Utility of the Technique during COVID-19 Pandemic. Medicines (Basel). 2021 Oct 19;8(10):60. doi: 10.3390/medicines8100060. PMID 34677489
- [Result] Kaya Ugur B, Pirbudak L, Ozturk E, Balat O, Ugur MG. Spinal versus general anesthesia in gynecologic laparoscopy: A prospective, randomized study. Turk J Obstet Gynecol. 2020 Sep;17(3):186-195. doi: 10.4274/tjod.galenos.2020.28928. Epub 2020 Oct 2. PMID 33072423